CLINICAL TRIAL: NCT04892979
Title: 3R Rehabilitation Management of COVID-19 Survivors Using Centre-based and Online-based Approaches
Brief Title: 3R Rehabilitation Management of COVID-19 Survivors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Pamela Youde Nethersole Eastern Hospital, Hong Kong (Unknown); Queen Elizabeth Hospital, Hong Kong (Other); Princess Margaret Hospital, Hong Kong (Other Government); Tuen Mun Hospital Hong Kong (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSEARS20200912001
Record Dates: First submitted 2021-03-01; First posted 2021-05-19 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-02

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Centre-based (Experimental): Centre-based exercise cardiopulmonary rehabilitation program for 6 weeks
  Interventions: Other: Cardiopulmonary exercise (centre-based)
- Online-based (Experimental): Online-based exercise cardiopulmonary rehabilitation program for 6 weeks
  Interventions: Other: Cardiopulmonary exercise (online-based)
- Combined (Experimental): Combined centre- and online-based exercise cardiopulmonary rehabilitation program for 6 weeks
  Interventions: Other: Cardiopulmonary exercise (centre-based); Other: Cardiopulmonary exercise (online-based)

INTERVENTIONS:
Other: Cardiopulmonary exercise (centre-based) — Depending on the preference of participants, they can either choose to join three 60-minute centre-based sessions plus two sessions of 30-minute home exercise per week, or two 60-minute centre-based sessions plus four sessions of 30-minute home exercise per week. Each session will include warm-up and cool-down exercises, aerobic exercises, and progressive strengthening exercises prescribed based on individual ability (Table 1). Aerobic exercises will be performed at 60-75% (up to 85% for fit individuals) of the predicted maximum heart rate. The respective rate of perceived exertion during exercise will be maintained between 4 and 6 out of 10 on the Borg CR scale [10], indicating moderate to strenuous exercise levels. Additionally, physiotherapists will provide education related to COVID-19, energy conservation, and stress management during the program.
  Arms: Centre-based; Combined
Other: Cardiopulmonary exercise (online-based) — Participants in the OBR group will attend one face-to-face session to learn how to use a mobile application (app) followed by 6 weeks of home exercises. The online treatments will be delivered via the Caspar Health e-system, a German-designed Internet-based system, is available for desktop PCs and as a mobile app for both iOS and Android smartphones. This system will enable patients to follow their therapists' treatment plans in an asynchronous manner. The OBR programme will last for 6 weeks. Participants will be instructed to perform 40 minutes of structured exercises 6 times per week. In the first week, six 40-minute online exercise sessions will be delivered through push notifications on the mobile app.
  Arms: Combined; Online-based

SUMMARY:
It is to explore the temporal relationships between physical fitness, cognitive, psychosocial functions, and health-related quality of life (HRQoL) in COVID-19 survivors over the first 15 months; and to determine the effects of centre-based (CBR), online-based cardiopulmonary rehabilitation (OBR), and combined centre- and online-based rehabilitation (COBR) on survivors with initially suboptimal pulmonary functions.

ELIGIBILITY:
Inclusion Criteria:

* COVID survivor at hospital discharge or 6-month post-disease onset
* Medically stable with an Abbreviated Mental Test (AMT) scores of > 6 out of 10

Exclusion Criteria:

* Having contraindications to exercise
* Physical Activity Readiness Questionnaire (PAR-Q) reveals unsafety
* Cannot understand Cantonese

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Fatigue measured by Fatigue Assessment Scale | 6 weeks after the start of intervention
  The Fatigue Assessment Scale is a 10-item scale evaluating symptoms of chronic fatigue.exercise test.
Fatigue measured by Fatigue Assessment Scale | Baseline
  The Fatigue Assessment Scale is a 10-item scale evaluating symptoms of chronic fatigue.exercise test.

SECONDARY OUTCOMES:
Muscle strength by 30-second double-leg sit-to-stand test (times) | Baseline
  Muscle strength will be assessed with the 30-second double-leg sit-to-stand test. If the participant can perform the 30-second single leg sit-to-stand test with pain or difficulty, they will be invited to complete 30-second single-leg sit-to-stand test. The number of completed repetitions will be counted.
Muscle strength by 30-second double-leg sit-to-stand test (times) | 6 weeks after the start of intervention
  Muscle strength will be assessed with the 30-second double-leg sit-to-stand test. If the participant can perform the 30-second single leg sit-to-stand test with pain or difficulty, they will be invited to complete 30-second single-leg sit-to-stand test. The number of completed repetitions will be counted.
Self-efficacy by 6-Item Chronic Disease Self-Efficacy scale | Baseline
  A six-item digital self-administered self-efficacy questionnaire will be used to evaluate patients' confidence in performing exercise, managing their own symptoms and emotions and completing their daily tasks.
Self-efficacy by 6-Item Chronic Disease Self-Efficacy scale | 6 weeks after the start of intervention
  A six-item digital self-administered self-efficacy questionnaire will be used to evaluate patients' confidence in performing exercise, managing their own symptoms and emotions and completing their daily tasks.
Self-perceived quality of life by The St. George's Respiratory Questionnaire-HK version | Baseline
  The St. George's Respiratory Questionnaire-HK version is a self-reported questionnaire. This 50-item disease specific questionnaire assesses 3 domains (symptoms, activity, and impacts).
Self-perceived quality of life by The St. George's Respiratory Questionnaire-HK version | 6 weeks after the start of intervention
  The St. George's Respiratory Questionnaire-HK version is a self-reported questionnaire. This 50-item disease specific questionnaire assesses 3 domains (symptoms, activity, and impacts).
Self-perceived quality of life by The Hong Kong Chinese version Short Form-36 | Baseline
  The Hong Kong Chinese version Short Form-36 is a concise 36-item health status questionnaire with good psychometric properties.
Self-perceived quality of life by The Hong Kong Chinese version Short Form-36 | 6 weeks after the start of intervention
  The Hong Kong Chinese version Short Form-36 is a concise 36-item health status questionnaire with good psychometric properties.
Cardiac output (L/min) | Baseline
  Non-invasive electrodes will be placed on the clavicle and lateral side of chest wall by a non-invasive measurement of cardiac output using the CardioScreen 1000 System. Non-invasive electrodes will be placed on the clavicle and lateral side of chest wall bilaterally
Cardiac output (L/min) | 6 weeks after the start of intervention
  Non-invasive electrodes will be placed on the clavicle and lateral side of chest wall by a non-invasive measurement of cardiac output using the CardioScreen 1000 System. Non-invasive electrodes will be placed on the clavicle and lateral side of chest wall bilaterally
Cardiac stroke volume (ml/m2) | Baseline
  Non-invasive electrodes will be placed on the clavicle and lateral side of chest wall by a non-invasive measurement of cardiac output using the CardioScreen 1000 System. Non-invasive electrodes will be placed on the clavicle and lateral side of chest wall bilaterally
Cardiac stroke volume (ml/m2) | 6 weeks after the start of intervention
  Non-invasive electrodes will be placed on the clavicle and lateral side of chest wall by a non-invasive measurement of cardiac output using the CardioScreen 1000 System. Non-invasive electrodes will be placed on the clavicle and lateral side of chest wall bilaterally
Forced expiratory volume in one second (l) | Baseline
  FEV1 is the volume of air that can forcibly be blown out in first 1 second, after full inspiration
Forced expiratory volume in one second (l) | 6 weeks after the start of intervention
  FEV1 is the volume of air that can forcibly be blown out in first 1 second, after full inspiration
Forced vital capacity (l) | Baseline
  Forced vital capacity (FVC) is the volume of air that can forcibly be blown out after full inspiration
Forced vital capacity (l) | 6 weeks after the start of intervention
  Forced vital capacity (FVC) is the volume of air that can forcibly be blown out after full inspiration
FEV1/FVC | Baseline
  Ratio of forced expiratory volume in one second and forced vital capacity
FEV1/FVC | 6 weeks after the start of intervention
  Ratio of forced expiratory volume in one second and forced vital capacity
Peak expiratory flow rate (l/s) | Baseline
  Peak expiratory flow (PEF) is the maximal flow (or speed) achieved during the maximally forced expiration initiated at full inspiration
Peak expiratory flow rate (l/s) | 6 weeks after the start of intervention
  Peak expiratory flow (PEF) is the maximal flow (or speed) achieved during the maximally forced expiration initiated at full inspiration
Exercise capacity (m) | Baseline
  Exercise capacity will be assessed by the 6-minute walk test (6MWT), a submaximal exercise test.
Exercise capacity (m) | 6 weeks after the start of intervention
  Exercise capacity will be assessed by the 6-minute walk test (6MWT), a submaximal exercise test.

CONTACTS AND LOCATIONS:
Overall Officials: Siu Ngor Fu, PhD, Principal Investigator — The Hong Kong Polytechnic University; Loletta Kit-ying So, MD, Principal Investigator — Pamela Youde Eastern Hospital
Locations (4):
- Hong Kong (4):
  - Pamela Youde Eastern Hospital, Hong Kong
  - Princess Margaret Hospital, Hong Kong
  - Queen Elizabeth Hospital, Hong Kong
  - Tuen Mun Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: No